CLINICAL TRIAL: NCT07189897
Title: An Open-label Pilot Study to Evaluate Medication Satisfaction With Apixaban Versus Enoxaparin for Thrombosis Prevention After Head and Neck Cancer Surgery
Brief Title: Apixaban or Enoxaparin After Head and Neck Cancer Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kiranya Arnold (Other)
Collaborators: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor-Investigator, Kiranya Arnold, Assistant Professor, State University of New York - Upstate Medical University
Organization: State University of New York - Upstate Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2225826-3
Record Dates: First submitted 2025-09-13; First posted 2025-09-24 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Venous Thromboembolism; Head and Neck Cancer
Keywords: surgery; apixaban; enoxaparin; thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Head and Neck Neoplasms; Thrombosis | interventions — Enoxaparin; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control: Enoxaparin (Active Comparator): 40 mg subcutaneous enoxaparin given once daily for DVT prevention.
  Interventions: Drug: Enoxaparin
- Experimental: Apixaban (Experimental): 2.5 mg oral apixaban given twice daily for DVT prevention.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Enoxaparin — For DVT prophylaxis
  Arms: Control: Enoxaparin
Drug: Apixaban — For DVT prophylaxis
  Arms: Experimental: Apixaban

SUMMARY:
The goal of this clinical trial is to learn if apixaban (a pill) is a safe and easier alternative to taking enoxaparin (a daily shot) to prevent blood clots after head and neck cancer surgery. It will also learn about side effects of both medicines.

The main questions it aims to answer are:

Can apixaban be used safely instead of enoxaparin to prevent blood clots after surgery? Do patients find apixaban easier or more satisfying to take than enoxaparin? How well do patients follow the treatment plan with each medicine?

Researchers will compare 2 groups:

One group will take apixaban (a pill taken twice a day) for 10 days after surgery.

The other group will take enoxaparin (a shot given once a day) for 10 days after surgery.

Participants will:

Take either apixaban or enoxaparin starting 12-24 hours after surgery, for 10 days total Keep a medication diary and bring back unused medicine so the study team can check adherence Complete short surveys about satisfaction with their medicine Have an ultrasound of their legs to check for blood clots 11-14 days after surgery Return for follow-up visits about 40 days and 80 days after surgery for safety checks

How long will participation last? About 4 months from surgery through the last follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Provide signed and dated informed consent.
* Be willing and able to comply with study procedures and follow-up.
* Be 18-89 years old (male or female).
* Have a negative pregnancy test within 24 hours before surgery (if woman of childbearing potential).
* Have biopsy-proven head and neck cancer, or a suspected cancer awaiting tissue diagnosis (can be confirmed by frozen section at surgery).
* Be scheduled for major inpatient or outpatient oncologic head and neck surgery (defined as >45 minutes operative time).
* Be an appropriate surgical candidate (adequate performance status).

Eligible diagnoses include (not limited to):

* Squamous cell carcinoma of oral cavity, hypopharynx, larynx, nasal cavity
* Malignancies from major salivary glands
* Non-melanoma skin cancers (squamous cell, basal cell, Merkel cell carcinoma)
* Unknown primary tumors of head and neck

Exclusion Criteria:

Participants cannot:

* Lack a tissue diagnosis of head and neck cancer during the study period.
* Have one of these conditions instead of eligible cancer: Benign disease; Primary thyroid cancer (lower VTE risk); Lymphoma (not primarily surgical); or Melanoma
* Fail to undergo definitive head and neck oncologic surgery (e.g., only diagnostic biopsy).
* Have surgery limited to tissue diagnosis only (e.g., direct laryngoscopy, excisional lymph node biopsy).
* Be unable (patient or caregiver) to administer the study drug.
* Have a positive pregnancy test on the day of surgery.
* Have a known history of prior DVT or PE (since extended anticoagulation would be indicated).
* Have hereditary or acquired bleeding/clotting disorders.
* Have severe renal impairment (CrCl <30 mL/min).
* Have conditions that, in the investigator's judgment, make study participation unsafe or confound results.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Study enrollment rate. | From study start until target enrollment is reached (up to 24 months).
  Enrollment rate will be calculated as the number of participants enrolled, divided by the number of eligible participants, multiplied by 100%.

SECONDARY OUTCOMES:
Medication satisfaction. | Assessed at Day 11-14 after completing 10 days of anticoagulant prophylaxis.
  Mean Anti-Clot Treatment Scale (ACTS) score. The ACTS comprises two primary subscales: ACTS Burdens and ACTS Benefits. The ACTS scores range from 12 to 60, but are often reverse-coded so that higher values indicate greater satisfaction. The ACTS Benefits scores range from 3 to 15, where higher scores reflect higher satisfaction.
Medication satisfaction. | Assessed at Day 11-14 after completing 10 days of anticoagulant prophylaxis.
  Mean Treatment Satisfaction Questionnaire for Medication (TSQM) - 1.4 score. TSQM 1.4 has four domains: Effectiveness, Side Effects, Convenience, and Global Satisfaction. Each domain is scored separately on a scale from 0 to 100, where higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No